CLINICAL TRIAL: NCT01333020
Title: A Pilot Study on the Effect of Protein Cross-linking on Gastric Layering and Emptying of a Food Emulsion
Brief Title: Cross-linked Emulsion Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IFR04/2010
Record Dates: First submitted 2011-04-08; First posted 2011-04-11 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Healthy Volunteers
Keywords: emulsion; protein; cross-linking; gastric emptying

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- transglutaminase cross-linking of emulsion (Experimental): The impact of enzyme cross linking of the protein stabilising the test emulsion on gastric emptying rate will be assessed. In this crossover study the subjects will also consume ( on a separate day)an emulsion of the same formulation but not cross-linked.
  Interventions: Other: cross-linking of an emulsion drink

INTERVENTIONS:
Other: cross-linking of an emulsion drink — This study will assess whether a subtle change in food structure (cross-linking of interfacial protein) can alter gastric emptying rate.

SUMMARY:
This comparative pilot study is designed to compare the rates of gastric emptying and by inference rates of digestion of two food emulsions. Two types of milk protein stabilised food emulsion will be compared, one standard emulsion preparation and one emulsion preparation cross-linked with microbial transglutaminase. The information from this study will then be compared to data on satiety and endocrine hormones from a parallel study undertaken in Finland using the same two meal formulations. The drinks will be labeled with a stable isotope of carbon and samples of breath collected every 20 minutes after consumption of the drink. This will allow gastric residence time to be calculated. The pilot will also fulfill two secondary objectives. At the same time as the breath samples are collected MRI scans of the upper abdomen will be made so that gastric volumes can be measured in order to compare the two methods of measuring gastric emptying rates. Additionally, samples of saliva will also be collected after every MRI scan for subsequent mass spectrometry analysis. These are to assess the efficacy of mass spectrometry analysis for detection of the presence of specific digestion related hormones such as ghrelin.

ELIGIBILITY:
Inclusion Criteria:

* Male (hormonal status of women would introduce more variation within small group)
* Age 20-50 years
* BMI 19-30
* Apparently healthy
* Normally eat lunch
* Willing to eat the "milkshake" style emulsion
* Provides written informed consent

Exclusion Criteria:

* You have an allergy or intolerance to rape seed oil, milk or milk proteins including lactose
* Smokers or smoked within the last year (smoking affects satiety/hunger)
* Diagnosed with any long term illness requiring active treatment e.g. diabetes, cancer, cardiovascular disease
* Have had surgery on the stomach or intestine or suffered from gastrointestinal disease, whether diagnosed or self reported
* A history of TB or hepatitis.
* Regular (more than once in 10 days) use of antacids, laxatives
* Diagnosis with any mouth, dental, throat or digestive problem that may affect normal eating and digestion of food.
* Take prescription medication for digestive or gastrointestinal conditions.
* Volunteers taking part in another study (other than a questionnaire based study).
* Blood pressure greater than 160/100 or less than 90/50 or 95/55 if symptomatic.
* Individuals with special dietary requirements (eg vegetarians)
* People with eating disorders (eg. anorexia, bulimia)
* If any of the clinical screening results are indicative of a health problem which would affect the volunteers well-being or which would affect the study data.
* Refusal to give permission to inform GP of participation in study
* Allergic to any of the constituents of the test meal
* Recent unexplained weight gain or loss
* History of back problems or any other condition which limit ability to repeatedly sit up and lie down
* Hiatus Hernia
* MRI scanning specific exclusion criteria

  * Cardiac pacemaker or artificial heart valve
  * Any surgery in the last 6 months
  * Aneurysm clips (metal clips from surgery)
  * Implant, pump or any medical device in the body (eg cochlear implant, neurostimulator, intra-ventricular shunt)
  * Worked with metals (using lathes or grinders) or sustained injury to eyes involving metal splinters or fillings
  * Have artificial eyes or limbs
  * Have been injured with shrapnel or bullets
  * Suffer from fits, blackouts or epilepsy
  * Claustrophobia sufferer

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2010-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Rate of gastric emptying by MRI | 20 minute intervals over 3 hours
  rate measured from MRI images of gastric contents

SECONDARY OUTCOMES:
Gastric emptying by C13 | every 20 minutes over 3 hours
  compare gastric emptying rates measured by MRI with those measured by 13C acetic acid breath tests.
mass spectrometry detection of GI tract hormones in saliva | every 20 minutes over 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alan R Mackie, PhD, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- IFR, Norwich, Norfolk, United Kingdom